CLINICAL TRIAL: NCT07136870
Title: Assessment of Wound Care Product Skin Adhesion
Acronym: SWAP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Essity Hygiene and Health AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: C3247 SWAP
Record Dates: First submitted 2025-08-15; First posted 2025-08-22 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Skin (FLACC Scores of Test Subjects) After Tape Removal
Keywords: Tape adhesion; Adhesion residues on skin; Tape removal sensation degree; medical tapes; wide area fixation; Post-Operative dressings

STUDY DESIGN:
Intervention Model Description: * Exploratory
  * Intra-individual comparison
  * Coded test samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group Tape wearing (Experimental): Sixteen samples of different test materials (medical tape) will be placed on the participant's upper and lower back. This ingle group acts as it's own control.
  Interventions: Device: Medical tape

INTERVENTIONS:
Device: Medical tape — The purpose of this exploratory study is to assess the adhesion to skin properties of test material samples over 24 hours to establish the peel-off measurement method at the new Essity study site. As the performance and safety of the tapes, WAFs and post-OPs in its intended use are not tested in the current study it is not considered a medical device study according to EU medical device regulation (MDR) 2017/745
  Other Names: Leukosilk tape; Fixomull stretch, wide area fixation tape; Fixomull skin sensitive, wide area fixation tape; Leukoplast tape; Fixomull transparent, wide area fixation tape; Leukopor tape; Leukomed, post-operative tape; Leukomed T skin sensitive, post-operative tape

SUMMARY:
The purpose of this exploratory study is to assess the adhesive forces to skin of samples over the period of 24 hours to establish the peel-off measurement method at the Essity study site.

DETAILED DESCRIPTION:
The main international standard for testing wound care products is EN 13726, which includes laboratory test methods for absorbency, fluid handling, breathability, adherence, and other physical characteristics of wound dressings. Different types of medical-grade adhesives are used, including rubber, acrylate, and silicone adhesives, each chosen based on the specific needs of the wound and the patient's skin. Proper application techniques are crucial for ensuring effective adhesion, such as ensuring the skin is clean and dry before applying the dressing, using side tabs to handle the dressing without touching the adhesive, and smoothing down the adhesive film to remove air bubbles.

Performance of all three product categories is reflected by general adhesion, e.g. to steel during quality control measurements and finally to skin when also considering the intended purpose of the product. Peel-off force measurement from tapes, WAFs and post-OPs applied to healthy skin are an established routine to compare different products and to test new adhesives or backings during new product development. Such measurements are conducted based on standardized peel-off methods which need to be established before running reliable quantitative measurements.

As the performance and safety of the tapes, WAFs and post-OPs in its intended use are not tested in the current study it is not considered a medical device study according to EU medical device regulation (MDR) 2017/745.

The samples will be investigated on female and male participants with healthy skin on the back (the application area). This assessment implies the determination of adhering properties to the skin, adhesive residues after removal of the samples as well as sensations during removal. Additionally, images of samples will be taken for documentation purposes.

ELIGIBILITY:
Inclusion Criteria:

* The participants must meet all of the following criteria to be eligible to participate in the investigation:

  1. Written informed consent to participate in the study.
  2. Willingness to actively participate in the study and to come to the scheduled visits.
  3. Female and/or male.
  4. From 18 to 70 years of age.
  5. Minimal hairiness on the back (the test area)

Exclusion Criteria:

* Participants meeting any of the following criteria will not be permitted to participate in the investigation:

  1. Female participants: Pregnancy or lactation.
  2. Drug or alcohol addiction.
  3. AIDS, HIV-positive or infectious hepatitis.
  4. Conditions which exclude a participation or might influence the test reaction/evaluation.
  5. Participation or being in the waiting period after participation in cosmetic and/or pharmaceutical studies pertaining to the test area.
  6. Cancer not being diagnosed as cured and requiring chemotherapy, irradiation and/or hormonal treatment within the last 2 years.
  7. Diabetes mellitus (type 1 and 2).
  8. One of the following illnesses with reduced physical capability/fitness: asthma (symptom-free allergic asthma is not an exclusion criterion), hypertension, cardiovascular diseases.
  9. Active skin disease at the test area.
  10. Documented allergies to dressings in particular with acrylates and natural rubber (latex).
  11. Wounds, moles, tattoos, scars, irritated skin at the test area that could influence the investigation.
  12. Any topical medication at the test area within the last 24 hours prior to the start of the study and/or throughout the entire course of the study.
  13. Application of cosmetics (e.g. creams, lotions, sunscreens) to the test area within the last 3 days prior to start of the study.
  14. Showering at the day of study start.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2026-02-11 (Estimated)

PRIMARY OUTCOMES:
Adhesion | After 24 hours of tape use
  Medical tape sample's adhesion force to skin measured in Newton-centimeter
Adhesive forces measured in N/cm | 1-2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Essity Study Site, Mölndal, VGR, Sweden

IPD SHARING:
Plan to Share IPD: No
IPD data will be only used internally by Essity and not be shared with other researchers.